CLINICAL TRIAL: NCT03375736
Title: Effect of Whole Body Vibration Therapy on Functional Abilities in Children and Young Adults With Moderate Severity of Cerebral Palsy- a Pilot Study
Brief Title: Whole Body Vibration for Children and Young Adults With Moderate Severity of Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YBW9
Record Dates: First submitted 2017-12-05; First posted 2017-12-18 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy
Keywords: whole body vibration; cerebral palsy; functional abilities; children; adults
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study participants would receive 4 weeks of whole body vibration therapy, 4 sessions per week for 18 minutes per session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Whole body vibration will be provided by an equipment, GalileoTM Med L Plus (Novotech Medical GmbH). The study participant will stand still on the vibration platform with both knees slightly flexed.
  Interventions: Device: whole body vibration

INTERVENTIONS:
Device: whole body vibration — The children and young adults will receive the WBVT when standing still on a vibration platform of 20 Hertz and a peak-to-peak amplitude of 2 mm: sessions will be 18 minutes in length, 4 days per week for 4 weeks. Assessments will be performed at baseline and at completion of the intervention to examine the functional abilities of these children and young adults. The vibration frequency, duration and amplitude will be progressively increased over 2 weeks to the maximum of 3 minutes of 20 Hz with a peak-to-peak amplitude of 2mm.

SUMMARY:
Osteopenia is common in children with cerebral palsy (CP) due to poor bone growth and muscle disuse and the problem extends to their adulthood. These children and young adults with CP, especially those with moderate physical disabilities, are unable to perform the required amount of exercise to improve their bone health as their typically developing counterparts. As a result, non-traumatic fractures and bone pain are common in individuals with moderate severity of CP. Whole body vibration therapy (WBVT) has been recently proven to improve bone health and muscle function in healthy adults and post-menopausal women. Among the research of the WBVT for children with CP, promising results have been shown on gross motor function, balance and muscle strength for children with mild disability. Among these published studies, the vibration protocols required the study participants to perform simple exercises on the vibration platform. Very limited studies have been conducted on children and young adults with moderate CP. At present, it is unknown if the effect of WBVT would be for this population group when compared with those with mild CP in terms of their gross motor function and balance, because the moderate group is greatly compromised in their mobility and extent of regular exercises when compared with the normal population and those with mild CP. In addition, it is unknown if static standing on the vibration platform would have similar effects on the gross motor function as doing simple exercises on the vibration platform. This pilot study aims to examine the effect of WBVT on children and young adults with moderate severity of CP. A convenience sample of 5 pre-puberty children aged between 6 to 14 years and 5 young adults aged between 18 to 40 years with moderate CP, i.e. Gross Motor Function Classification System, GMFCS level III or IV, will be recruited to systematically investigate the effects of WBVT on their functional abilities.

DETAILED DESCRIPTION:
Osteopenia is common in children with cerebral palsy (CP) due to poor bone growth and muscle disuse and the problem extends to their adulthood. These children and young adults with CP, especially those with moderate physical disabilities, are unable to perform the required amount of exercise to improve their bone health as their typically developing counterparts. It has been demonstrated that strong bones or good bone health are related to muscle contractions during normal movements and regular exercises. As a result, non-traumatic fractures and bone pain are common in individuals with moderate severity of CP. Whole body vibration therapy (WBVT) has been recently proven to improve bone health and muscle function in healthy adults and post-menopausal women. It has been postulated that the vibration can stimulate the muscle spindles and elicit consistent muscle contractions. This would be a great advantage to the individuals with physical disabilities, who have limited movements and control in their body and prevent them to perform regular exercises as the normal individuals. Among the research of the WBVT for children with CP, promising results have been shown on gross motor function, balance and muscle strength for children with mild disability. Among these published studies, the vibration protocols required the study participants to perform simple exercises on the vibration platform. Very limited studies have been conducted on children and young adults with moderate CP. At present, it is unknown if the effect of WBVT on this population group would be similar to those with mild CP in terms of their gross motor function and balance, because the moderate group is greatly compromised in their mobility and extent of regular exercises when compared with the normal population and those with mild CP. It is also unknown if static standing on the vibration platform would have similar effects on the gross motor function as doing simple exercises on the vibration platform.

This pilot study aims to examine the effect of WBVT on children and young adults with moderate severity of CP. A convenience sample of 5 pre-puberty children aged between 6 to 14 years and 5 young adults aged between 18 to 40 years with moderate CP, i.e. Gross Motor Function Classification System, GMFCS level III or IV, will be recruited to systematically investigate the effects of WBVT on their functional abilities. Individuals with GMFCS level III mobilise with hand-held mobility devices such as crutches or walking frames. Individuals of levels IV have very limited functional mobility and are mostly limited to an indoor environment.

The children and young adults will receive the WBVT when standing still on a vibration platform of 20 Hertz and a peak-to-peak amplitude of 2 mm: sessions will be 18 minutes in length, 4 days per week for 4 weeks. Assessments will be performed at baseline and at completion of the intervention to examine the changes in the functional abilities of these children and young adults. The vibration frequency, duration and amplitude will be progressively increased over 2 weeks to the maximum of 3 minutes of 20 Hz with a peak-to-peak amplitude of 2mm and remain the same for the rest of the 2 weeks.

The outcomes of this pilot study will show if this intervention is beneficial for children and young adults with moderate CP with respect to their functional abilities, and if there may be any related practical issues of this intervention to this population group. The outcomes also provide preliminary evidence to clinicians if this intervention is effective to improve functional abilities of children and young adults with moderate severity of CP and provide preliminary data to calculate sample sizes for future studies.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of cerebral palsy with Gross Motor Function Classification System, GMFCS level III or IV
* able to stand on a vibration platform independently or by holding rails on their own
* able to follow simple instructions

Exclusion Criteria:

* a history of fracture within 8 weeks of enrolment of the present study and acute thrombosis, muscle or tendon inflammation, renal stones, discopathy or arthritis as reported by their parent/ guardian.
* behavioral problems that prevent them to follow simple instructions
* females who are pregnant
* any metal implant

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Changes in Gross Motor Function Measure (GMFM-66) item set | at 0 and 4 weeks
  to assess changes in the gross motor function of study participants

SECONDARY OUTCOMES:
Changes in 2-minute walk test (2MWT) | at 0 and 4 weeks
  to assess changes in submaximal exercise capacity of the study participants by measuring the distance covered in 2 minutes using a distance-measuring trundle wheel
Changes in Chinese version of the Pediatric Evaluation of Disability Inventory (PEDI) | at 0 and 4 weeks
  to assess changes in the functional capacities in the domains of daily activities, mobility and social/cognitive function
Changes in Timed up and go test | at 0 and 4 weeks
  to assess changes in the balance and functional mobility of the study participants by measuring the time used to perform this test
Parental/ participant questionnaire | at 4 weeks
  to record satisfaction (0 means not satisfied and 10 as extreme satisfied) and any comments on the intervention regime as reported by the study participants and/or by their carers' proxy
Visual analogue scale | after each intervention session up to 4 weeks
  to assess discomfort (0 means no discomfort and 10 as extreme discomfort), if any, associated with the intervention as reported by the study participants and/or by their carers' proxy

CONTACTS AND LOCATIONS:
Overall Officials: Tamis W Pin, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Anonymous individual and group data would be submitted for publication.

REFERENCES:
- [Result] Sheridan KJ. Osteoporosis in adults with cerebral palsy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:38-51. doi: 10.1111/j.1469-8749.2009.03432.x. PMID 19740209
- [Result] Rauch F. Vibration therapy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:166-8. doi: 10.1111/j.1469-8749.2009.03418.x. PMID 19740225
- [Result] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus Mallen JA. Effect of whole-body vibration therapy on health-related physical fitness in children and adolescents with disabilities: a systematic review. J Adolesc Health. 2014 Apr;54(4):385-96. doi: 10.1016/j.jadohealth.2013.11.001. Epub 2014 Jan 1. PMID 24388109
- [Result] Saquetto M, Carvalho V, Silva C, Conceicao C, Gomes-Neto M. The effects of whole body vibration on mobility and balance in children with cerebral palsy: a systematic review with meta-analysis. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):137-44. PMID 26032205
- [Result] Houlihan CM, Stevenson RD. Bone density in cerebral palsy. Phys Med Rehabil Clin N Am. 2009 Aug;20(3):493-508. doi: 10.1016/j.pmr.2009.04.004. PMID 19643349
- [Result] van den Berg-Emons HJ, Saris WH, de Barbanson DC, Westerterp KR, Huson A, van Baak MA. Daily physical activity of schoolchildren with spastic diplegia and of healthy control subjects. J Pediatr. 1995 Oct;127(4):578-84. doi: 10.1016/s0022-3476(95)70115-x. PMID 7562279
- [Result] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Result] Mergler S, Evenhuis HM, Boot AM, De Man SA, Bindels-De Heus KG, Huijbers WA, Penning C. Epidemiology of low bone mineral density and fractures in children with severe cerebral palsy: a systematic review. Dev Med Child Neurol. 2009 Oct;51(10):773-8. doi: 10.1111/j.1469-8749.2009.03384.x. Epub 2009 Jul 8. PMID 19614941
- [Result] Cheng HY, Ju YY, Chen CL, Chuang LL, Cheng CH. Effects of whole body vibration on spasticity and lower extremity function in children with cerebral palsy. Hum Mov Sci. 2015 Feb;39:65-72. doi: 10.1016/j.humov.2014.11.003. Epub 2014 Nov 24. PMID 25461434
- [Result] Kilebrant S, Braathen G, Emilsson R, Glansen U, Soderpalm AC, Zetterlund B, Westerberg B, Magnusson P, Swolin-Eide D. Whole-body vibration therapy in children with severe motor disabilities. J Rehabil Med. 2015 Mar;47(3):223-8. doi: 10.2340/16501977-1921. PMID 25613047
- [Result] Unger M, Jelsma J, Stark C. Effect of a trunk-targeted intervention using vibration on posture and gait in children with spastic type cerebral palsy: a randomized control trial. Dev Neurorehabil. 2013;16(2):79-88. doi: 10.3109/17518423.2012.715313. PMID 23477461
- [Result] Ahlborg L, Andersson C, Julin P. Whole-body vibration training compared with resistance training: effect on spasticity, muscle strength and motor performance in adults with cerebral palsy. J Rehabil Med. 2006 Sep;38(5):302-8. doi: 10.1080/16501970600680262. PMID 16931460
- [Result] Dickin DC, Faust KA, Wang H, Frame J. The acute effects of whole-body vibration on gait parameters in adults with cerebral palsy. J Musculoskelet Neuronal Interact. 2013 Mar;13(1):19-26. PMID 23445911
- [Result] Gusso S, Munns CF, Colle P, Derraik JG, Biggs JB, Cutfield WS, Hofman PL. Effects of whole-body vibration training on physical function, bone and muscle mass in adolescents and young adults with cerebral palsy. Sci Rep. 2016 Mar 3;6:22518. doi: 10.1038/srep22518. PMID 26936535
- [Result] Russell DJ, Avery LM, Walter SD, Hanna SE, Bartlett DJ, Rosenbaum PL, Palisano RJ, Gorter JW. Development and validation of item sets to improve efficiency of administration of the 66-item Gross Motor Function Measure in children with cerebral palsy. Dev Med Child Neurol. 2010 Feb;52(2):e48-54. doi: 10.1111/j.1469-8749.2009.03481.x. Epub 2009 Oct 7. PMID 19811516
- [Result] Pin TW. Psychometric properties of 2-minute walk test: a systematic review. Arch Phys Med Rehabil. 2014 Sep;95(9):1759-75. doi: 10.1016/j.apmr.2014.03.034. Epub 2014 May 9. PMID 24814460
- [Result] Chen KL, Hsieh CL, Sheu CF, Hu FC, Tseng MH. Reliability and validity of a Chinese version of the Pediatric Evaluation of Disability Inventory in children with cerebral palsy. J Rehabil Med. 2009 Mar;41(4):273-8. doi: 10.2340/16501977-0319. PMID 19247548
- [Result] Williams EN, Carroll SG, Reddihough DS, Phillips BA, Galea MP. Investigation of the timed 'up & go' test in children. Dev Med Child Neurol. 2005 Aug;47(8):518-24. doi: 10.1017/s0012162205001027. PMID 16108451
- [Derived] Pin TW, Butler PB, Purves S. Use of whole body vibration therapy in individuals with moderate severity of cerebral palsy- a feasibility study. BMC Neurol. 2019 May 1;19(1):80. doi: 10.1186/s12883-019-1307-5. PMID 31043157

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT03375736/Prot_SAP_000.pdf